CLINICAL TRIAL: NCT05087888
Title: Investigation of Serial Advanced Magnetic Resonance Imaging (MRI) and Biofluid Biomarkers Predictive of Neurocognitive Decline Following Brain Radiation
Brief Title: MRI and Blood Biomarkers for the Prediction of Neurocognitive Decline Following Brain Radiation
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: PA18-0719; NCI-2021-09725 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PA18-0719 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-10-05; First posted 2021-10-21 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Brain Neoplasm
MeSH Terms: conditions — Brain Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood

GROUPS / COHORTS (1):
- Observational (MRI, questionnaire, blood collection): Patients undergo multiparametric MRI with contrast at baseline, 3 weeks during radiotherapy, and at 1, 3, 6, 12, and 24 months post-radiotherapy. Patients undergo multiparametric MRI without contrast at 1, 2, 4, 5, and 6 weeks during radiotherapy. Patients may undergo functional MRI at baseline and 6 months post-radiotherapy. Patients also complete questionnaires and undergo collection of blood samples at baseline, weekly through week 6 during radiotherapy, and at 1, 3, 6, 12, and 24 months post radiotherapy.
  Interventions: Procedure: Biospecimen Collection; Procedure: Magnetic Resonance Imaging; Procedure: Multiparametric Magnetic Resonance Imaging; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection
Procedure: Magnetic Resonance Imaging — Undergo functional MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Multiparametric Magnetic Resonance Imaging — Undergo multiparametric MRI
  Other Names: MP-MRI; mpMRI; Multi-parametric MRI; Multiparametric MRI
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This study determines whether non-invasive evaluation using repeated magnetic resonance imaging (MRI) scans and repeated blood biomarker measurements can be used to predict changes in a person's mental functions that result from radiation exposure to the brain. This study may let researchers monitor patient responses to treatment and the disease better and possibly make changes to patient treatment, if needed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To describe changes of image features on conventional T1- and T2- weighted imaging, and quantitative changes on multiparametric MRI including apparent diffusion coefficient (ADC), fractional anisotropy (FA), relative cerebral blood volume (rCBV), fractional volume of the extravascular, extracellular space (ve) and Ktrans (transfer constant that characterizes the diffusive transport of low-molecular weight gadolinium across the capillary endothelium) associated with neurocognitive changes following radiation.

SECONDARY OBJECTIVES:

I. To identify biofluid biomarkers at baseline and dynamics of biomarkers after radiation exposure that are associated with neurocognitive changes.

II. To model a composite early biomarker (baseline or within 3 weeks of the start of radiotherapy) that incorporates the most promising imaging and biofluid biomarkers to predict for later neurocognitive decline.

III. To evaluate the relationship between the delivered radiation dosimetry to brain subregions and patterns of neurocognitive decline in order to inform potential subregions of focus for future pre-clinical and clinical investigation.

IV. To evaluate the relationship between quantitative changes on multiparametric MRI including apparent diffusion coefficient (ADC), fractional anisotropy (FA), relative cerebral blood volume (rCBV), fractional volume of the extravascular, extracellular space (ve) and Ktrans (transfer constant that characterizes the diffusive transport of low-molecular weight gadolinium across the capillary endothelium) with radiation dosimetry.

EXPLORATORY OBJECTIVE:

I. To explore changes on advanced MR measurements of structural connectomics, functional connectomics, working memory network, cerebrovascular reactivity (CVR), cerebral blood flow (CBF) and brain metabolism associated with neurocognitive changes following radiation.

OUTLINE:

Patients undergo multiparametric MRI with contrast at baseline, 3 weeks during radiotherapy, and at 1, 3, 6, 12, and 24 months post-radiotherapy. Patients undergo multiparametric MRI without contrast at 1, 2, 4, 5, and 6 weeks during radiotherapy. Patients may undergo functional MRI at baseline and 6 months post-radiotherapy. Patients also complete questionnaires and undergo collection of blood samples at baseline, weekly through week 6 during radiotherapy, and at 1, 3, 6, 12, and 24 months post radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be age >= 18 years
* Patients must be planned for fractionated radiotherapy that will be delivered over at least 5 weeks and that will expose the brain to radiation
* Patients must have Karnofsky performance status (KPS) >= 80
* Patients must be able to obtain an MRI scan with gadolinium contrast
* Female patients of childbearing age must not be pregnant as determined with a serum beta human chorionic gonadotropin (HCG) no greater than 14 days prior to study registration, or breast-feeding. (The exclusion is made because gadolinium may be teratogenic in pregnancy). Pregnancy tests are part of standard of care routine if a patient is receiving radiation treatment
* Patient must be fluent enough in English to complete neurocognitive testing
* Education of >= 12 years (high school graduate or equivalent) by patient self-report
* Patient is able to complete an in-person and electronic neurocognitive assessments (i.e. is alert and has the ability to comprehend and complete the assessments)
* Patient has no history of psychiatric or medical conditions that would result in an inability to complete serial neurocognitive tests, severe claustrophobia, prior cerebrovascular event(s), degenerative neurological diagnoses (e.g., dementia, Parkinson's, multiple sclerosis [MS]) or severe psychiatric illness (e.g., schizophrenia) that may impact neurocognitive and imaging assessments

Exclusion Criteria:

* Previous brain radiation without comprehensive dosimetry records
* Concurrent chemotherapy
* Psychiatric or medical conditions that would result in inability to complete serial neurocognitive tests
* Severe claustrophobia requiring sedative medications for the MRI
* Prior cerebrovascular event(s) or degenerative neurological diagnoses (e.g., dementia, Parkinson's, MS)
* Contraindication to gadolinium-based contrast administration for MRI (i.e. allergy to gadolinium or severe chronic kidney disease defined by estimated glomerular filtration rate [eGFR] < 30 mL/min/1.73 m^2, as per institutional policy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing central nervous system (CNS) or head and neck (H&N) radiotherapy with radiation exposure to the brain to investigate the pattern of neurocognitive changes in relation to brain dosimetry and associated imaging and biofluid biomarkers predictive of neurocognitive outcomes
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
To describe changes of image features on conventional T1- and T2- weighted imaging, and quantitative changes on the multipara metric MRI. | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Chung, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M.D. Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2023-09-29): https://cdn.clinicaltrials.gov/large-docs/88/NCT05087888/ICF_000.pdf